CLINICAL TRIAL: NCT07208175
Title: Effectiveness of Ultrasound-guided Peripheral Intravenous Catheter (EUPIC) Insertion Versus Traditional (Touch and Feel) Insertion Approaches by Oncology Nurses. A Mixed-methods Randomized Controlled Trial (RCT).
Brief Title: Effectiveness of Ultrasound-Guided Versus Traditional IV Insertion by Oncology Nurses in Adult Population Recieving Systemic Anti-cancer Therapy.
Acronym: EUPIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Galway (Other)
Responsible Party: Principal Investigator, Caitriona Duggan, PhD candidate, University of Galway
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Ref: C.A 3374; CNRA21DUG. (Other Grant/Funding Number: Irish Cancer Society)
Record Dates: First submitted 2025-09-27; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-Guided Peripheral Intravenous Catheter (PIVC) Insertion (Experimental): Ultrasound-Guided Peripheral Intravenous Catheter (PIVC) Insertion Participants randomized to this arm will undergo PIVC insertion performed by trained oncology nurses using real-time ultrasound guidance. The ultrasound device will be used to assess and select a suitable vein, guide needle advancement, and confirm catheter placement. This approach is designed to improve first-time insertion success, preserve vein health, and reduce insertion-related complications compared to the traditional touch-and-feel technique.
  Interventions: Other: Ultrasound-Guided Peripheral Intravenous Catheter Insertion
- Traditional (Touch-and-Feel) Peripheral Intravenous Catheter (PIVC) Insertion (Active Comparator): Traditional (Touch-and-Feel) Peripheral Intravenous Catheter (PIVC) Insertion Participants randomized to this arm will receive PIVC insertion performed by oncology nurses using the standard landmark technique. This method relies on visual inspection and palpation of the vein to guide catheter placement, without the use of ultrasound. It reflects current routine clinical practice for establishing intravenous access in oncology patients.
  Interventions: Other: Traditional Peripheral Intravenous Catheter Insertion

INTERVENTIONS:
Other: Ultrasound-Guided Peripheral Intravenous Catheter Insertion — In this arm, PIVC insertion is performed by oncology nurses who have completed a structured ultrasound training program. Nurses use real-time ultrasound imaging to identify and select a suitable vein, guide the advancement of the catheter, and confirm placement. This method contrasts with the standard touch-and-feel approach by incorporating ultrasound technology and specialized nurse training to improve first-time insertion success and reduce complications.
  Arms: Ultrasound-Guided Peripheral Intravenous Catheter (PIVC) Insertion
Other: Traditional Peripheral Intravenous Catheter Insertion — PIVC insertion performed by oncology nurses using the conventional touch-and-feel landmark technique, relying on visual inspection and palpation of veins. Represents current standard clinical practice in oncology.
  Arms: Traditional (Touch-and-Feel) Peripheral Intravenous Catheter (PIVC) Insertion

SUMMARY:
What is this study about? This study is comparing two different methods nurses use to place an intravenous (IV) drip, which is needed for many cancer treatments.

Traditional method: The nurse finds a vein by touch and sight.

Ultrasound-guided method: The nurse uses a small, handheld ultrasound scanner to see the vein under the skin to help guide the needle.

Why is it important? Sometimes it can take more than one attempt to get an IV drip in place, which can be uncomfortable. For cancer patients, whose veins can be more fragile, this is a common challenge. This research will help us find out if using ultrasound helps get the IV in successfully on the first try more often, which can make the treatment experience better.

What does participation involve? If you choose to take part, you will be randomly assigned (like a coin toss) to have your IV placed with either the traditional method or the ultrasound method. The research team will then collect some information about the IV placement. Your participation is entirely voluntary and will not affect your standard medical care.

DETAILED DESCRIPTION:
Title

Effectiveness of Ultrasound-guided Peripheral Intravenous Catheter (EUPIC) insertion versus traditional (touch and feel) insertion approaches by oncology nurses: A mixed-methods Randomized Controlled Trial (RCT).

Background and Rationale

Peripheral intravenous catheters (PIVCs) are a cornerstone of cancer treatment, allowing the delivery of systemic anti-cancer therapies (SACT) such as chemotherapy, immunotherapy, targeted agents, and supportive drugs. However, first-time insertion success (FTIS) is often suboptimal, particularly in oncology patients with difficult intravenous access (DIVA) due to prior vein damage, dehydration, obesity, or treatment-induced changes.

The traditional landmark method (sight and palpation) remains the dominant approach but is associated with high variability in FTIS and frequent multiple attempts. These failures result in patient discomfort, anxiety, treatment delays, and increased healthcare costs.

Ultrasound-guided (USG) insertion has demonstrated improved outcomes in general hospital populations. Still, evidence in oncology is limited, with a Cochrane review finding low-certainty evidence and highlighting the need for high-quality randomized controlled trials in this specific group.

Given the vulnerability of cancer patients and the importance of vein preservation for long-term therapy, this study investigates whether USG PIVC insertion, performed by trained oncology nurses, improves outcomes compared to the traditional method.

Objectives

Primary Objective:

To determine if ultrasound-guided PIVC insertion improves first-time insertion success compared with the traditional touch-and-feel technique in adult cancer patients undergoing SACT.

Secondary Objectives:

Evaluate catheter longevity and dwell time.

Assess patient-reported outcomes (pain, anxiety, satisfaction, quality of life).

Document complications (e.g., phlebitis, occlusion, infiltration, dislodgement, bloodstream infection).

Measure procedural efficiency (time to insertion).

Assess the impact of ultrasound training on oncology nurses' competence and confidence.

Explore patients' and clinicians' experiences of both approaches through qualitative interviews.

Study Design

Type: Mixed-methods, two-arm randomized controlled trial (RCT) with an embedded qualitative component.

Sites: Three oncology units across the HSE West and North West (designated cancer centre, nurse-led oncology day unit, community oncology satellite).

Sample Size: 98 participants (49 per group). Calculation assumes FTIS of 0.70 (traditional) vs. 0.90 (USG), with 80% power at α = 0.05.

Recruitment: Multi-site, opportunistic during routine cancer care. Patients will be approached before treatment, given information, and allowed time to consent.

Eligibility Criteria

Inclusion:

Adults ≥18 years.

Diagnosis of cancer requiring SACT.

Requiring PIVC insertion.

Exclusion:

<18 years.

Inability to provide informed consent.

Unable to cooperate with study procedures.

Interventions Control Arm - Traditional Technique

Carried out by oncology nurses competent in PIVC placement.

Relies on anatomical palpation and visual assessment to guide insertion.

Intervention Arm - Ultrasound-Guided Technique

Nurses trained at the University of Galway in USG vascular access.

Real-time ultrasound used to assess veins, guide needle insertion, and confirm placement.

Training includes task analysis, supervised practice, and competency assessment.

Outcomes Primary Outcome

First-time insertion success (FTIS): Successful placement of PIVC on the first attempt.

Secondary Outcomes

Catheter failure rates before completion of therapy (dislodgement, occlusion, infiltration, phlebitis, infection).

Procedure time - time from request to successful insertion.

Device dwell time - duration from insertion to removal.

Referral for alternative vascular access devices (VADs).

Nurse competence and confidence - assessed via surveys and interviews pre/post training.

Patient-reported pain - measured using Numerical Rating Scale (0-10).

Patient anxiety and quality of life - Beck Anxiety Inventory, EQ-5D.

Patient and clinician qualitative experiences - semi-structured interviews exploring perceptions of comfort, pain, anxiety, and procedural acceptability.

Data Collection

Baseline: Demographics, diagnosis, vein assessment (palpation and ultrasound metrics), and DIVA status.

During insertion: Device type and size, location, attempts, procedural time, FTIS.

Follow-up: Daily monitoring (inpatients) or routine checks (outpatients) for complications, dwell time, premature removal.

Patient-reported outcomes: Pain, anxiety, QoL questionnaires.

Qualitative: Audio-recorded interviews transcribed verbatim and analysed thematically (Braun & Clarke framework).

Randomization and Allocation

1:1 ratio using computer-generated permuted blocks.

Stratified randomization ensures balanced allocation across cancer subgroups.

Blinding: Not feasible for patients or nurses due to intervention nature.

Statistical Analysis

Primary outcome: Proportion of FTIS compared using chi-square tests and logistic regression adjusting for baseline covariates (age, sex, site).

Secondary outcomes:

Time-to-event outcomes (Kaplan-Meier survival analysis, Cox proportional hazards models).

Comparisons of continuous variables (parametric/non-parametric tests).

Confidence intervals reported; significance set at p < 0.05.

Qualitative data: Systematic coding in NVivo, thematic analysis (familiarization, coding, theme development, interpretation).

Safety and Monitoring

Data Safety Monitoring Committee (DSMC): Independent panel (oncologist, anaesthetist, trialist). Reviews SAEs and progress.

Serious Adverse Events (SAEs): Reported immediately to DSMC.

Auditing: Continuous internal monitoring; no external audit planned given low-risk nature.

Ethics and Governance

Ethical approval: Clinical Research Ethics Committee, Galway University Hospital.

Consent: Obtained by research team, with assurance of voluntary participation and withdrawal rights.

Confidentiality: Data anonymized, stored securely in REDCap, compliant with GDPR.

Amendments: Substantial changes require REC approval; updates shared with registry and stakeholders.

Dissemination

Results will be published in peer-reviewed open-access journals (e.g., Trials).

Findings will be presented at national and international oncology and nursing conferences.

Results will be shared with participants, clinical teams, and patient advocacy groups.

Trial registration and summary results will be updated on ClinicalTrials.gov.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 years or older.

Diagnosed with cancer (all cancer sites eligible).

Scheduled to receive systemic anti-cancer therapy (SACT) such as chemotherapy, immunotherapy, or targeted therapies.

Requiring peripheral intravenous catheter (PIVC) insertion for treatment.

Exclusion Criteria:

* Patients younger than 18 years.

Individuals unable to provide informed consent.

Individuals unable to cooperate with study procedures (e.g., cognitive or physical limitations preventing adherence).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-10-20 (Estimated); Primary Completion 2025-12-23 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
First-time insertion success (FTIS) of peripheral intravenous catheter | At time of PIVC insertion (single insertion episode; assessed immediately following the procedure)
  Proportion of participants with successful peripheral intravenous catheter placement on the first skin-puncture attempt. Success is defined as successful cannulation on the first needle puncture with confirmation of a functioning PIVC by (1) visible/aspirable blood return and (2) ability to flush and infuse a standard 10 mL saline bolus without resistance or infiltration. The outcome is recorded as a binary variable (Yes/No) on the case report form by the treating/research nurse immediately after the procedure and used to calculate the percentage of FTIS per arm.

CONTACTS AND LOCATIONS:
Overall Officials: Caitriona Duggan, Principal Investigator — University of Galway

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results reported in future publications will be made available to other researchers upon reasonable request to the corresponding author. Data sharing will require approval from the trial sponsor and a signed data access agreement. Data will only be shared for ethically approved research purposes and in compliance with GDPR and institutional policies.
Supporting Information: Study Protocol
Time Frame: De-identified individual participant data (IPD) will be made available after publication of the primary trial results. Data will remain available for up to 7 years following publication.
Access Criteria: De-identified individual participant data (IPD) and supporting documents (including the study protocol, statistical analysis plan, and informed consent form) will be made available to qualified researchers affiliated with academic institutions, healthcare organizations, or non-commercial research groups. Access will be granted for scientifically and ethically approved research projects.
  Researchers must submit a written request to the corresponding author outlining the study objectives, methods, and intended use of the data. Requests will be reviewed by the trial sponsor and principal investigators. Upon approval, a data access agreement must be signed before IPD is shared. Data will be provided in secure electronic format in compliance with GDPR and institutional policies.